CLINICAL TRIAL: NCT06257264
Title: A Phase 1a/1b Study of BG-68501, a Selective CDK2 Inhibitor, in Participants With Advanced Solid Tumors
Brief Title: A Study to Examine the Safety of Different Doses of BG-68501 Given to Participants With Advanced-Stage Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BG-68501-101; CTR20243059 (Registry Identifier: ChinaDrugTrials.org); 2024-517324-19-00 (EU CTIS Number)
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Small Cell Lung Cancer; Ovarian Cancer; Gastric Cancer; Hormone-receptor-positive Breast Cancer; Hormone Receptor Positive HER-2 Negative Breast Cancer; Advanced Solid Tumor; Endometrial Cancer; Prostate Cancer; TNBC - Triple-Negative Breast Cancer; GastroEsophageal Cancer; Bladder Cancer
Keywords: breast cancer; small cell lung cancer; ovarian cancer; gastric cancer; cdk2 inhibitor; BG-68501; HR+ HER2- breast cancer; endometrial cancer; prostate cancer; BGB-43395; bladder cancer; urothelial cancer; gastroesophageal cancer; cdk4 inhibitor; fulvestrant
MeSH Terms: conditions — Breast Neoplasms; Small Cell Lung Carcinoma; Ovarian Neoplasms; Stomach Neoplasms; Endometrial Neoplasms; Prostatic Neoplasms; Triple Negative Breast Neoplasms; Urinary Bladder Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1 Part A: Dose Escalation and Safety Expansion (BG-68501 Monotherapy) (Experimental): Sequential cohorts of increasing dose levels of BG-68501 will be evaluated as monotherapy.
  Interventions: Drug: BG-68501
- Part 1 Part B: Dose Escalation (BG-68501 + Fulvestrant) (Experimental): Sequential cohorts of increasing dose levels of BG-68501 will be evaluated in combination with fulvestrant.
  Interventions: Drug: BG-68501; Drug: Fulvestrant
- Part 1 Part C: Dose Escalation and Safety Expansion (BG-68501 + Fulvestrant + BGB-43395) (Experimental): Sequential cohorts of increasing dose levels of BG-68501 will be evaluated in combination with fulvestrant and BGB-43395.
  Interventions: Drug: BG-68501; Drug: Fulvestrant; Drug: BGB-43395
- Part 1: Food Effect Evaluation (Experimental): Participants will receive BG-68501 at a dose level that is determined safe and tolerable to evaluate food effect. Food effect may also be evaluated for BG-68501 in combination with fulvestrant.
  Interventions: Drug: BG-68501; Drug: Fulvestrant
- Part 2: Dose Expansion (Experimental): The RFDE for BG-68501 (as monotherapy and in combination with fulvestrant and BGB-43395) from Part 1 will be evaluated in selected tumor cohorts.
  Interventions: Drug: BG-68501; Drug: Fulvestrant; Drug: BGB-43395

INTERVENTIONS:
Drug: BG-68501 — Planned doses administered orally.
Drug: Fulvestrant — Standard dose administered via intramuscular injection.
  Arms: Part 1 Part B: Dose Escalation (BG-68501 + Fulvestrant); Part 1 Part C: Dose Escalation and Safety Expansion (BG-68501 + Fulvestrant + BGB-43395); Part 1: Food Effect Evaluation; Part 2: Dose Expansion
Drug: BGB-43395 — Planned doses administered orally.
  Arms: Part 1 Part C: Dose Escalation and Safety Expansion (BG-68501 + Fulvestrant + BGB-43395); Part 2: Dose Expansion

SUMMARY:
This study is a first-in-human (FIH), Phase 1a/1b study of BG-68501, a cyclin-dependent kinase-2 inhibitor (CDK2i), to assess the safety, tolerability, pharmacokinetics (PK), pharmacodynamics, and preliminary antitumor activity of BG-68501 in participants with advanced, nonresectable, or metastatic solid tumors as monotherapy and in combination with fulvestrant with or without BGB-43395, a selective CDK4 inhibitor, in adults with hormone receptor positive (HR+)/human epidermal growth factor receptor 2 negative (HER2-) breast cancer (BC). The study will also identify a recommended dose for expansion (RDFE) for BG-68501 as monotherapy and in combination for subsequent disease directed studies.

The study will be conducted in 2 parts: Part 1 (dose escalation and safety expansion, including evaluation of food effect) and Part 2 (dose expansion).

ELIGIBILITY:
Part 1 (Dose Escalation) Inclusion Criteria:

* Monotherapy Cohorts: Participants with histologically or cytologically confirmed advanced or metastatic solid tumors potentially associated with CDK2 dependency including HR+/HER2- breast cancer, platinum refractory or resistant serous ovarian cancer (PROC), endometrial cancer, and others. Prior available standard-of-care systemic therapies for advanced or metastatic disease are required. The requirements for enrollment into a food effect evaluation cohort are the same as the monotherapy cohorts with the exception that participants with gastric cancer and gastroesophageal adenocarcinoma are excluded.
* Combination Cohorts (BG-68501 with fulvestrant with or without BGB-43395): Enrollment is restricted to only participants with HR+/HER2- BC. In regions where approved and available, participants must have received one or more lines of treatment for advanced/metastatic disease as well as prior endocrine therapy and a CDK4/6 inhibitor in either the adjuvant or advanced/metastatic setting. If applicable, the requirements for enrollment into a food effect evaluation cohort are the same as the combination cohorts.

Part 1 (Safety Expansion) and Part 2 (Dose Expansion) Inclusion Criteria:

* Participants with advanced, non-resectable, or metastatic HR+/HER2- BC or PROC, including fallopian tube or primary peritoneal cancer.
* PROC participants must have received:

  * ≥ 1 line of platinum-containing chemotherapy for advanced disease.
  * ≤ 4 prior therapeutic regimens in the advanced/metastatic setting.
* HR+/HER2- BC:

  * Participants enrolled in regions where CDK4/6 inhibitors are approved and available must have received ≥ 1 line of therapy including endocrine therapy and a CDK4/6 inhibitor. Participants can have received up to 2 lines of prior cytotoxic chemotherapy or ADC treatments for advanced disease.

General Inclusion Criteria:

* Female participants with advanced or metastatic HR+/HER2- BC will be required to have ovarian function suppression using gonadotropin hormone-releasing hormone (GnRH) agonists (such as goserelin) or be postmenopausal.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1.
* Adequate organ function.
* For dose escalation, participants with advanced solid tumors other than HR+/HER2- BC must have measurable disease per RECIST 1.1. Participants with HR+/HER2- BC with bone-only disease are eligible for dose escalation only. For safety expansion and dose expansion, all participants must have ≥1 measurable lesion per RECIST v 1.1.

General Exclusion Criteria:

* For all cohorts: Prior therapy selectively targeting CDK2 inhibition.
* For triple combination cohorts: Prior therapy targeting CDK2 or selectively targeting CDK4. Prior CDK4/6 inhibitor therapy is permitted and required in local regions where it is approved and available.
* Known leptomeningeal disease or uncontrolled, untreated brain metastasis. Participants with a history of treated central nervous system (CNS) metastases may be eligible if they meet additional criteria.
* Any malignancy ≤ 3 years before the first dose of study treatment(s) except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated with curative intent (eg, resected basal or squamous cell skin cancer, superficial bladder cancer, treated papillary thyroid carcinoma, or carcinoma in situ of the cervix or breast).
* Uncontrolled diabetes.
* Infection requiring systemic antibacterial, antifungal, or antiviral therapy antiviral therapy ≤ 28 days before the first dose of study drug(s), or symptomatic COVID-19 infection.
* Active hepatitis B infection or active hepatitis C infection.
* Any major surgical procedure ≤ 28 days before the first dose of study treatment(s).
* Prior allogeneic stem cell transplantation, or organ transplantation.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From the first dose of study drug(s) to 30 days after the last dose; approximately 6-12 months
  Number of participants with treatment-emergent AEs and SAEs.
Part 1: Maximum Tolerated Dose (MTD) or Maximum Administered Dose (MAD) of BG-68501 | Up to approximately 24 months
  MTD is defined as the highest dose evaluated for which estimated toxicity rate is the closest to the target toxicity rate. MAD is defined as the highest dose administered if MTD is not reached.
Part 1: Recommended dose(s) for Expansion (RDFE) of BG-68501 monotherapy in participants with solid tumors | Up to approximately 24 months
  RDFE of BG-68501 alone will be determined based upon the MTD or MAD.
Part 1: RDFE of BG-68501 in combination with fulvestrant and BGB-43395 in participants with HR+/HER2- BC | Up to approximately 24 months
  RDFE of BG-68501 in combination with fulvestrant and BGB-43395 will be determined based upon the MTD or MAD.
Part 2: Objective Response Rate (ORR) | Up to approximately 20 months
  ORR is defined as the percentage of participants with best overall response of complete response (CR) or partial response (PR). CR and PR that is confirmed by repeat assessments, as assessed by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

SECONDARY OUTCOMES:
Part 1: ORR | Up to approximately 20 months
  ORR is defined as the percentage of participants with best overall response of CR or PR. CR and PR that is confirmed by repeat assessments, as assessed by the investigator using RECIST v1.1.
Part 2: Number of participants with AEs and SAEs | From the first dose of study drug(s) to 30 days after the last dose; approximately 6-12 months
  Number of participants with AEs and SAEs, including findings from physical examinations, electrocardiograms (ECGs), and laboratory assessments.
Parts 1 and 2: Duration of Response (DOR) | Up to approximately 20 months
  DOR is defined as the time from the first confirmed objective response by the investigator using RECIST v1.1 until the first documentation of disease progression after treatment initiation or death, whichever comes first.
Parts 1 and 2: Time to Response (TTR) | Up to approximately 20 months
  TTR is defined as the time from the treatment initiation to the first determination of overall response by the investigator using RECIST v1.1.
Parts 1 and 2: Disease Control Rate (DCR) | Up to approximately 20 months
  DCR is defined as the percentage of participants with the best overall response, of a CR, PR, and stable disease assessed by the investigator using RECIST v1.1.
Parts 1 and 2: Clinical Benefit Rate (CBR) | Up to approximately 20 months
  CBR is defined as the percentage of participants with best overall response of confirmed CR, PR, or stable disease lasting ≥ 24 weeks assessed by the investigator using RECIST v1.1.
Part 1: Maximum observed plasma concentration (Cmax) for BG-68501 and BGB-43395 | 2 times in the first 2 months
Part 1: Observed plasma trough concentration (Ctrough) for BG-68501 and BGB-43395 | 5 times in the first 2 months
Part 1: Area under the concentration-time curve (AUC) for BG-68501 and BGB-43395 | 2 times in the first 2 months
Part 1: Half-life (t1/2) for BG-68501 and BGB-43395 | 2 times in the first 2 months
Part 2: Plasma concentrations for BG-68501 and BGB-43395 | 5 times in approximately 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (24):
- United States (6):
  - Hoag Memorial Presbyterian, Newport Beach, California
  - Florida Cancer Specialists and Research Institute, Lake Mary, Florida
  - Washington University School of Medicine, St Louis, Missouri
  - Titan Health Partners Llc Dba Astera Cancer Care, East Brunswick, New Jersey
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Mary Crowley Cancer Research, Dallas, Texas
- Australia (7):
  - Blacktown Cancer and Haematology Centre, Blacktown, New South Wales
  - Saint Vincents Hospital Sydney, Darlinghurst, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Genesiscare North Shore, St Leonards, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Cancer Research South Australia, Adelaide, South Australia
  - Monash Health, Clayton, Victoria
- China (7):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Sun Yat Sen Memorial Hospital, Sun Yat Sen University (South), Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Hunan Cancer Hospital, Changsha, Hunan
  - Shengjing Hospital Affiliated of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi
- Israel (2):
  - Rambam Health Care Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
- The Institute of Oncology, Arensia Exploratory Medicine, Chisinau, Moldova
- Auckland City Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/